CLINICAL TRIAL: NCT02062255
Title: A Phase 0, Investigator Initiated Study, Evaluating the Impact of COX2 Inhibition on Human Sera Biomarkers From Obese Subjects
Brief Title: Impact of COX2 on Sera Biomarkers From Obese Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Andrew Brenner, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CTRC 13-0041; HSC20130426H (Other: UTHSCSA IRB)
Record Dates: First submitted 2013-12-09; First posted 2014-02-13 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer Survivors
Keywords: Asprin; Omega-3 Free Fatty Acids; Obesity; COX-2 inhibitor
MeSH Terms: conditions — Obesity | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aspirin (Active Comparator): Twenty eight enteric coated 81mg Aspirin tablets will be dispensed for daily oral dosing, to be taken with a meal at the same time of day.
  Interventions: Drug: Aspirin
- Omega-3 Free Fatty Acids (Active Comparator): Three hundred thirty-six gelatin coated 450 mg capsules containing approximately 180 mg of EPA and 135 mg of DHA will be dispensed. Patients are to take 12 capsules daily with meals, either once daily (12 capsules with one meal) or divided twice daily (e.g., six with breakfast and six with dinner).
  Interventions: Dietary Supplement: Omega 3 FFA
- Aspirin & Omega-3 FFAs (Active Comparator): Aspirin (81 mg po daily) to be taken simultaneously with Omega-3 Free Fatty Acids (1500mg of docosahexaoic acid (DHA) and 2500mg eicosapentanoic acid (EPA) given daily.
  Interventions: Drug: Aspirin; Dietary Supplement: Omega 3 FFA

INTERVENTIONS:
Drug: Aspirin
  Arms: Aspirin; Aspirin & Omega-3 FFAs
Dietary Supplement: Omega 3 FFA
  Arms: Aspirin & Omega-3 FFAs; Omega-3 Free Fatty Acids

SUMMARY:
Obesity promotes worse outcome for post-menopausal breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Post-menopausal as confirmed by medical history
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee

Exclusion Criteria:

* Evidence of active cancer (patients with a prior history of malignancy are encouraged to participate, but due to cytokine levels associated with malignancy there must be no evidence of disease)
* Cachexia
* Active systemic illness (infection including viral illnesses such as Hepatitis and HIV)
* Chronic use of aspirin of omega-3 free fatty acid supplementation within the last 60 days (defined as greater than or equal to 7 consecutive days)
* Known hypersensitivity to aspirin and/or omega-3 fatty acids
* Actively receiving a physician-directed regimen of aspirin and/or receiving herapeutic/prophylactic anticoagulation
* Any aspirin or omega-3 free fatty acid supplementation within the last 14 days
* Subjects who are pregnant
* History of medical noncompliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Biomarker levels | 29 days
  Blood levels of Prostaglandin E2, aromatase, pro-inflammatory cytokines, steroids, and lipids will be measured pre and post treatment.

SECONDARY OUTCOMES:
BMI | 29 Days
  Correlation for body mass index impact on response to COX2 inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brenner, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas, United States